CLINICAL TRIAL: NCT04731298
Title: An Open Label, Single Arm, Multicentre, Proof of Concept, Phase 2 Study to Investigate the Pharmacokinetics, Pharmacodynamics and Assess the Efficacy and Safety to Support Dose Selection of Emapalumab in Pre-empting Graft Failure in Patients at High Risk After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Study to Investigate the Pharmacokinetics, Pharmacodynamics and Assess the Efficacy and Safety to Support Dose Selection of Emapalumab in Pre-empting Graft Failure in Patients at High Risk After HSCT.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision related to Business Priorities, Assessment of Development Options
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: PRA Health Sciences (Industry); Cytel Inc. (Industry); Q2 Solutions (Industry); ABF Pharmaceutical Services GmbH (Industry); Cromsource (Industry); BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NI-0501-12
Record Dates: First submitted 2020-11-13; First posted 2021-01-29 (Actual); Results first posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Graft Failure
Keywords: HSCT; allo-HSCT; Graft failure; emapalumab; interferon gamma; CXCL9
MeSH Terms: interventions — Emapalumab

STUDY DESIGN:
Intervention Model Description: Sequential dose cohorts. The first cohort of patients will receive a first emapalumab infusion of 6 mg/kg at TD0, followed by a second infusion at 3 mg/kg after 3 days. Subsequent infusions of 3 mg/kg will be every 3 or 4 days from previous dose until dose 15 or until engraftment. A maximum of 2 additional cohorts may be added to allow dosing regimen adaptation based on the PK/PD data observed from the previous cohort(s).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emapalumab (Experimental): The first cohort of patients will receive a first infusion of 6 mg/kg at TD0, followed by a second infusion at 3 mg/kg after 3 days (treatment day 3 - TD3). Subsequent infusions of 3 mg/kg will be every 3 or 4 days from previous dose until dose 15 or until engraftment.
  A maximum of 2 additional cohorts may be added to allow dosing regimen adaptation based on the PK/PD data observed from the previous cohort(s). Efficacy and safety data will also be considered before adding additional cohorts.
  Interventions: Drug: Emapalumab

INTERVENTIONS:
Drug: Emapalumab — Emapalumab is a fully human immunoglobulin G1 (IgG1) anti-IFNγ monoclonal antibody that binds to and neutralizes IFNγ. Emapalumab binds to both soluble and receptor (IFNγR1)-bound forms of IFNγ.
  Emapalumab is in development for treatment of primary and secondary HLH. The benefit expected from the targeted neutralization of IFNγ by emapalumab has been validated by the recent FDA approval of emapalumab for treatment of patients with pHLH who have refractory, recurrent or progressive disease or intolerance with conventional HLH therapy. The safety profile has been assessed as acceptable.
  Emapalumab will be administered by intravenous infusion over 1 to 2 hours, depending on the volume of the infusion. The first infusion must be performed within 12 hours after CXCL9 levels have been measured above defined threshold. Treatment will last until maximum dose 15 (up to 56 days) or until evidence of engraftment, whichever comes first.
  Other Names: Gamifant®; NI-0501

SUMMARY:
This study is designed as an open-label, single arm, proof of concept study in order to determine the appropriate emapalumab dosing regimen neutralizing IFNγ in patients at risk of GF. Patients presenting CXCL9 levels above a defined threshold and other clinical criteria will be eligible to receive emapalumab.

Both children and adults, with malignant and non-malignant underlying diseases, receiving allo-HSCT who are at high risk of GF as defined in the inclusion criteria will be included in the study. The main objective of the study is to determine the appropriate emapalumab dose regimen neutralizing interferon gamma (IFNγ) activity to pre-empt graft failure post allo-HSCT in a population with various underlying diseases and at high risk of graft failure (GF).

Maximum 3 cohorts are foreseen to determine the appropriate dose regimen to pre-emptively treat patients at risk of primary GF.

Emapalumab will be administered by IV infusion and treatment will last up to 56 days (15 infusions) or until evidence of engraftment.

The study is expected to last approximately 3 years from screening to the last follow-up phone call for each patient.

DETAILED DESCRIPTION:
This study is designed as an open-label, single arm, proof of concept study in order to determine the appropriate emapalumab dosing regimen neutralizing IFNγ in patients at risk of GF. Patients presenting CXCL9 levels above a defined threshold and other clinical criteria will be eligible to receive emapalumab.

Both children and adults, with malignant and non-malignant underlying diseases, receiving allo-HSCT who are at high risk of GF as defined in the inclusion criteria will be included in the study. The main objective of the study will be to determine the appropriate emapalumab dose regimen neutralizing interferon gamma (IFNγ) activity to pre-empt graft failure post allo-HSCT in a population with various underlying diseases and at high risk of graft failure (GF).

Maximum 3 cohorts are foreseen to determine the appropriate dose regimen to pre-emptively treat patients at risk of primary GF.

Emapalumab will be administered by IV infusion over 1 to 2 hours depending on the volume of the infusion. Treatment will last up to 56 days (15 infusions) or until evidence of engraftment.

The study is comprised of the following study periods: screening (Day -21 to Day -8), allogeneic HSCT Day 0, monitoring period for primary GF (Day 1 up to Day 42), extended monitoring for secondary GF (up to Day 98), treatment period (up to 56 days) and follow-up period of 3 years after HSCT.

The main objective of this proof of concept study is:

• To determine the appropriate emapalumab dose regimen neutralizing interferon gamma (IFNγ) activity to pre-empt graft failure post allogeneic hematopoietic stem cell transplantation (HSCT) in a population with various underlying diseases and at high risk of graft failure (GF)

The following objectives will support the dose selection:

* To describe the Pharmacokinetic (PK) and Pharmacodynamic (PD) profiles of emapalumab post allogeneic HSCT (allo-HSCT)
* To assess the efficacy of emapalumab to pre-empt GF post allo-HSCT
* To assess the safety of emapalumab to pre-empt GF post allo-HSCT
* To assess the immunogenicity of emapalumab post allo-HSCT

Exploratory objectives will be:

• To evaluate further data on the correlation between relevant biomarkers including C-X-C motif chemokine ligand 9 (CXCL9) levels and the risk of GF post allo-HSCT in a population with various underlying diseases and at high risk of GF also in the context of development of a diagnostic test.

The study is expected to last approximately 3 years from screening to the last follow-up phone call for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed by the patient (as required by law) or by the patient's legally authorized representative(s) with the assent of patients who are legally capable of providing it, as applicable
2. Recipients of allogeneic Hematopoietic Stem Cell Transplantation (HSCT) and at high risk of graft failure (GF) based on at least one of the following criteria:

   * Receiving reduced intensity conditioning (RIC) or non-myeloablative conditioning (NMA) combined with a non-malignant disease or with a graft from Bone Marrow (BM)
   * Ex vivo T cell depleted graft
   * Graft from mismatched unrelated or haploidentical donor
   * Graft from Umbilical Cord Blood (UCB)
3. Patients requiring allo-HSCT with the following underlying diseases:

   * Malignant disease with high risk of GF, i.e. Acute Myeloid Leukemia (AML) and Acute Lymphoblastic Leukemia (ALL) with primary induction failure, second partial remission or relapse; Chronic Myeloid Leukemia (CML) in blastic phase (circulating blast or blast above 5% in biopsy); Non Hodgkin and Hodgkin Lymphoma and multiple myeloma with primary induction failure, second partial remission or relapse, myelodysplastic syndromes (MDS) and myeloproliferative disorders (MPD) with splenomegaly, myelofibrosis with portal hypertension pre-transplant, MDS/MPD overlap syndromes
   * Non-malignant hematological diseases (e.g. autoimmune and metabolic disorders, aplastic anemia, Sickle cell anemia, Fanconi anemia, Diamond-Blackfan anemia, thalassemia, osteopetrosis, Wiskott-Aldrich syndrome, severe combined immunodeficiency, Hemophagocytic lymphohistiocytosis and other immunoregulatory disorders)
4. Male and female patients
5. Children aged at least 1 year and adults. Once the appropriate dose has been determined in one of the three cohorts and safety has been assessed by the Independent Data Monitoring Committee (IDMC), children less than 1 year old may be included in the study.
6. Females of child-bearing potential, defined as all women physiologically capable of becoming pregnant, require use of highly effective contraceptive measures from screening until 6 months after the last study drug administration

Exclusion Criteria:

1. Pregnant (or planning to become pregnant) or lactating female patients
2. Body weight < 3 kg
3. Underlying malignant disease with Karnofsky/Lansky performance status equal or less than 40 or an Eastern Cooperative Oncology Group (ECOG) performance status equal or less than 3
4. Patients presenting CXCL9 levels 10 times above the upper limit of the 95% interval (CI) of the normal range (reported in the CXCL9 assay laboratory manual) within 24 hours prior to HSCT
5. Clinically manifested infections caused by typical and atypical Mycobacteria, Salmonella, Histoplasma capsulatum and Herpes Zoster on the day of HSCT
6. Active or clinical suspicion of latent tuberculosis
7. Concomitant diseases that in the opinion of the Investigator may interfere with the assessment of emapalumab safety or efficacy
8. Receipt of a Bacille Calmette-Guerin (BCG) vaccine within 3 months prior to HSCT
9. Receipt of a live or attenuated live (other than BCG) vaccine within 6 weeks prior to HSCT
10. Current or scheduled administration of therapies known to potentially trigger a cytokine release syndrome within 21 days from HSCT.
11. Patients having received IFNγ during the last 2 weeks prior to HSCT and/or who require treatment with IFNγ.
12. Patients having received emapalumab during the last 6 months prior to HSCT, unless it is known that emapalumab is no longer detectable.
13. Patients having received kinase inhibitors (Janus kinase inhibitors [JAKi] or bruton tyrosine kinase inhibitors [BTKi]) one week (or 5 half-lives whichever is greater) prior to HSCT.
14. Intolerance to antimicrobial and virus infection prophylaxis.
15. Hypersensitivity to emapalumab or any of the excipients.
16. Ongoing participation in an interventional trial or administration of any investigational drug (within 3 half-lives of the investigational drug) with the exception of interventional trials involving supportive care such as probiotics or antiemetics, graft manipulation, or use of new combinations or new dosing of conventional therapies for conditioning and prophylaxis pre-HSCT.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsila Zuckerman, Dr, Principal Investigator — The Rambam Academic Hospital; Henrique Bittencourt, Dr, Principal Investigator — St. Justine's Hospital; Polina Stepensky, Dr, Principal Investigator — Hadassah Hebrew University; Ashvind Prabahran, Dr, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Richard Mitchell, Dr, Principal Investigator — Kids Cancer Centre Sydney Children's Hospital
Locations (5):
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne
  - Kids Cancer Centre Sydney Children's Hospital, Randwick
- CHU Sainte-Justine, Montreal, Quebec, Canada
- Israel (2):
  - The Rambam Academic Hospital, Haifa
  - Hadassah Hebrew University, Jerusalem

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One site was activated which screened a total of 3 subjects (2 enrolled; 1 screen failure). First and last subjects were enrolled 25May2021 and 07Oct2021 respectively.
Groups:
- Emapalumab Treated: Patients treated with emapalumab (i.e. patients who met the protocol requirements for initiating emapalumab treatment)
- Non-emapalumab Treated: Patients not treated with emapalumab (i.e.patients who did not meet the protocol requirements for initiating emapalumab treatment)
Period: Allogeneic HSCT (Day 0)
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0
Period: Monitoring - Primary GF (Day 1 to 42)
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0
Period: Monitoring - Secondary GF (Up to Day 98)
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0
Period: Follow-up (3 Years From HSCT)
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2
Not completed — Early termination of study. | 0 | 2

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in the emapalumab arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Emapalumab Treated | Non-emapalumab Treated | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 2 | 2
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 2 | 2
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada |  | 2 | 2
Underlying disease: Aplastic anemia [Count of Participants; unit: Participants] |  | 2 | 2
Graft - Type of conditioning [Count of Participants; unit: Participants] — Engraftment was defined as absolute neutrophils count (ANC) >= 500 cells/microliter (mcL) for 3 consecutive measures and donor chimerism above 60% or ANC >= 500 cells/mcL for 3 consecutive measures and 2 consecutive measures of donor chimerism above 60% or 7 days of platelets above 20000 cells/mcL without transfusion.
  Participants
    Non myeloablative regimen (NMA) |  | 1 | 1
    Reduced Intensity Conditioning (RIC) |  | 1 | 1
Graft - Source of stem cells [Count of Participants; unit: Participants]
  Peripheral blood stem cell (PBSC) |  | 1 | 1
  Bone marrow (BM) |  | 1 | 1
Graft - Donor type [Count of Participants; unit: Participants]
  Matched unrelated donor |  | 1 | 1
  Mismatched unrelated donor |  | 1 | 1
Number of transplanted cells [Median (Full Range); unit: million cells] |  | 290.9 [83.5 to 498.3] | 290.9 [83.5 to 498.3]
ABO incompatibility [Count of Participants; unit: Participants]
  Major |  | 1 | 1
  No incompatibility |  | 1 | 1
Mean CXCL9 concentration (prior to HSCT) [Median (Full Range); unit: pg/mL] |  | 203.50 [181.00 to 226] | 203.5 [181 to 226]

OUTCOME MEASURES:

1. Primary Outcome: CXCL9 in Serum
Description: Serum concentration of C-X-C Motif Chemokine Ligand 9 (CXCL9)
Time Frame: From start of treatment to EoS Visit, up to 34 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Primary Graft Failure (GF)
Description: Number of participants with primary graft failure (GF)
Time Frame: From Hematopoietic stem-cell transplantation (HSCT) [Day 0] up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Secondary GF
Description: Number of participants with secondary GF
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Free & Total Interferon Gamma (IFNγ) in Serum
Description: Serum concentration of free and total Interferon gamma (IFNγ)
Time Frame: From start of treatment to EoS Visit, up to 34 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Emapalumab in Serum - Peak
Description: Peak emapalumab serum concentration
Time Frame: From start of treatment to EoS, up to 34 weeks
Population: No patients enrolled in the emapalumab arm.
Groups:
- Emapalumab: Patients treated with emapalumab (i.e. patients who met the protocol requirements for initiating emapalumab treatment)
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Ctrough (Emapalumab)
Description: Concentration just before administration
Time Frame: From start of treatment to EoS, up to 34 weeks
Population: No patients enrolled in the emapalumab arm.
Arm/Group | Emapalumab Treated
Number analyzed (Participants) | 0

7. Secondary Outcome: Exploratory Biomarkers: Ferritin
Description: Ferritin - serum concentration
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: ADA and nAbs
Description: Number of participants developing antibodies against emapalumab (antidrug antibodies [ADA]) and Neutralizing antibodies (nAb)
Time Frame: From Start of treatment until EoS, up to 34 weeks
Population: No patients enrolled in the emapalumab arm.
Arm/Group | Emapalumab Treated
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Mixed Donor Chimerism <10% and <20%
Description: Based on unselected leukocytes and based on sorted T cells
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No patients enrolled in the emapalumab arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

10. Secondary Outcome: Number of Participants Receiving Thrombopoietic Agents, Stem Cell Boost, Donor Lymphocyte Infusion (DLI)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants Receiving a Second Allogeneic HSCT
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Poor Graft Function
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Event Free Engraftment
Description: defined as absence of GF or graft support
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No patients enrolled in the emapalumab arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 2
Participants | 0 | 2

14. Secondary Outcome: Number of Participants With Acute and/or Chronic Mild to Severe Graft Versus Host Disease (GvHD)
Description: (grade I to IV)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No patients enrolled in the emapalumab arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 2
Participants | 0 | 1

15. Secondary Outcome: Biomarker Levels, in Particular IFNy and CXCL9, as Predictors of Primary and/or Secondary Graft Failure or Acute and/or Chronic GvHD
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Engraftment Syndrome
Description: Number of participants with engraftment syndrome
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No patients enrolled in the emapalumab arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 2
Participants | 0 | 1

17. Secondary Outcome: Number of Participants With Endothelial Complications
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Number of Participants With Relapse, Defined as Cumulative Incidence of Reoccurring Underlying Disease
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Survival Rate
Description: Number of patients alive at the end of study.
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No patients enrolled in the emapalumab arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 2
Participants |  | 2

20. Secondary Outcome: Change in Body Temperature
Description: Change from baseline in body temperature
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change in Heart Rate
Description: Change from baseline in heart rate
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change in Blood Pressure
Description: Change from baseline systolic and diastolic blood pressure
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change in Body Weight
Description: Change from baseline in body weight
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Change in Hematology: Red Blood Cells (RBC)
Description: Change from baseline in Hematology: red blood cells (RBC)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Change in Hematology: Hematocrit
Description: Change from baseline in Hematology: hematocrit
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Change in Hematology: Hemoglobin
Description: Change from baseline in Hematology: hemoglobin
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Change in Hematology: Platelets
Description: Change from baseline in Hematology: platelets
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Change in Hematology: White Blood Cells (WBC)
Description: Change from baseline in Hematology: white blood cells (WBC)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Change in Hematology Differential: Lymphocytes
Description: Change from baseline in Hematology differential: lymphocytes
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Change in Hematology Differential: Monocytes
Description: Change from baseline in Hematology differential: monocytes
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Change in Hematology Differential: Neutrophils
Description: Change from baseline in Hematology differential: neutrophils
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Change in Biochemistry: Ferritin
Description: Change from baseline in Biochemistry: Ferritin
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Change in Biochemistry: Glucose
Description: Change from baseline in Biochemistry: Glucose
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Change in Biochemistry: C-reactive Protein
Description: Change from baseline in Biochemistry: C-reactive protein
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Change in Biochemistry: Sodium
Description: Change from baseline in Biochemistry: Sodium
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Change in Biochemistry: Potassium
Description: Change from baseline in Biochemistry: Potassium
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Change in Biochemistry: Chloride
Description: Change from baseline in Biochemistry: Chloride
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Change in Biochemistry: Calcium
Description: Change from baseline in Biochemistry: Calcium
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Change in Biochemistry: Magnesium
Description: Change from baseline in Biochemistry: Magnesium
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Change in Biochemistry: Phosphate
Description: Change from baseline in Biochemistry: Phosphate
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Change in Biochemistry: Aspartate Aminotransferase (AST)
Description: Change from baseline in Biochemistry: Aspartate aminotransferase (AST)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Change in Biochemistry: Alanine Aminotransferase (ALT)
Description: Change from baseline in Biochemistry: alanine aminotransferase (ALT)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Change in Biochemistry: Gamma-glutamyl Transpeptidase (γGT)
Description: Change from baseline in Biochemistry: gamma-glutamyl transpeptidase (γGT)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Change in Biochemistry: Alkaline Phosphatase (ALP)
Description: Change from baseline in Biochemistry: alkaline phosphatase (ALP)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Change in Biochemistry: Lactate Dehydrogenase (LDH)
Description: Change from baseline in Biochemistry: lactate dehydrogenase (LDH)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Change in Biochemistry: Bilirubin
Description: Change from baseline in Biochemistry: bilirubin (total, direct and indirect)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Change in Biochemistry: Triglycerides
Description: Change from baseline in Biochemistry: triglycerides
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Change in Biochemistry: Cholesterol
Description: Change from baseline in Biochemistry: cholesterol (total and high-density lipoprotein [HDL])
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Change in Biochemistry: Albumin
Description: Change from baseline in Biochemistry: Albumin
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Change in Biochemistry: Creatinine
Description: Change from baseline in Biochemistry: Creatinine
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Change in Biochemistry: Urea
Description: Change from baseline in Biochemistry: Urea
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Activated Partial Thromboplastin (aPTT)
Description: Change from baseline in Coagulation: activated partial thromboplastin (aPTT)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

53. Secondary Outcome: Prothrombin Time (PT)
Description: Change from baseline in Coagulation: prothrombin time (PT)
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Change in Urinalysis: Glucose
Description: Change from baseline in Urinalysis: Glucose
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Change in Urinalysis: Blood
Description: Change from baseline in Urinalysis: Blood
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Change in Urinalysis: Protein
Description: Change from baseline in Urinalysis: Protein
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Change in Urinalysis: Leucocytes
Description: Change from baseline in Urinalysis: Leucocytes
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Change in Urinalysis: Ketones
Description: Change from baseline in Urinalysis: Ketones
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

59. Secondary Outcome: Change in Urinalysis: pH
Description: Change from baseline in Urinalysis: pH
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

60. Secondary Outcome: Change in Urinalysis: Specific Gravity
Description: Change from baseline in Urinalysis: specific gravity
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

61. Secondary Outcome: Number of Subjects With Change in Donor Chimerism
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No patients enrolled in the emapalumab arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 2
Participants
  Change = 100% | 0 | 2
  Change < 100% | 0 | 0

62. Secondary Outcome: Change in HLA Antibodies
Description: Change from baseline in HLA antibodies against donor cells
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

63. Secondary Outcome: Change From Baseline in Minimal Residual Disease (MRD)
Description: Only in patients presenting malignant disease
Time Frame: From HSCT (Day 0) up to study termination, approximately 46 weeks
Population: No efficacy data was collected since no subject received study treatment.
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to study termination, approximately 46 weeks
Description: No patients were enrolled in the emapalumab arm.
Groups:
- Emapalumab Treated: Patients treated with emapalumab
Arm/Group | Emapalumab Treated | Non-emapalumab Treated
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emapalumab Treated (N=0) | Non-emapalumab Treated (N=2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | 2 (2)
Flushing (Vascular disorders) | NA | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | NA | 2 (3)
Constipation (Gastrointestinal disorders) | NA | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | NA | 1 (1)
Bradycardia (Cardiac disorders) | NA | 1 (1)
Hypertension (Vascular disorders) | NA | 2 (2)
Hepatic enzyme increased (Investigations) | NA | 1 (1)
Chills (General disorders) | NA | 1 (1)
Pyrexia (General disorders) | NA | 2 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | NA | 2 (2)
Sepsis (Infections and infestations) | NA | 1 (1)
Headache (Nervous system disorders) | NA | 2 (2)
Nausea (Gastrointestinal disorders) | NA | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | NA | 1 (1)
Abdominal pain (Gastrointestinal disorders) | NA | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | NA | 1 (2)
Nephropathy toxic (Renal and urinary disorders) | NA | 1 (1)
Graft versus host disease in skin (Immune system disorders) | NA | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | NA | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | 1 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | NA | 1 (2)
Hypervolaemia (Metabolism and nutrition disorders) | NA | 1 (3)
Mucosal inflammation (General disorders) | NA | 1 (1)
Insomnia (Psychiatric disorders) | NA | 1 (1)
Perineal abscess (Infections and infestations) | NA | 1 (2)
Engraftment syndrome (Immune system disorders) | NA | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | NA | 1 (2)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | NA | 1 (1)
Salmonella test positive (Investigations) | NA | 1 (1)
Injection site pain (General disorders) | NA | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | NA | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | NA | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | NA | 1 (1)
Allergy to immunoglobulin therapy (Immune system disorders) | NA | 1 (1)
Ingrown toe nail (Skin and subcutaneous tissue disorders) | NA | 1 (1)
Chemokine increase (Investigations) | NA | 1 (1)
Drug hypersensitivity (Immune system disorders) | NA | 1 (1)
Non-cardiac chest pain (General disorders) | NA | 1 (1)
Diarrhoea (Gastrointestinal disorders) | NA | 1 (1)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated with only 2 patients enrolled. Both patients were in the non-emapalumab treated arm, i.e. no patients received study treatment (emapalumab). Consequently, the majority of analyses were not performed and no conclusion on the efficacy of emapalumab on this patient population could be drawn from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT04731298/Prot_SAP_000.pdf